CLINICAL TRIAL: NCT01801280
Title: Pharmacokinetic Cross-over Study to Evaluate the Influence of Pantoprazole on MPA Bioavailability Administered as Mycophenolate Mofetil and Enteric Coated Mycophenolate Sodium in Maintenance Renal Transplant Patients
Brief Title: Influence of Pantoprazole on the Bioavailability of MMF and EC-MPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Klemens Budde (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Klemens Budde, Professor Dr Klemens Budde, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CERL 080A DE 20 T; 2010-021275-92 (EudraCT Number)
Record Dates: First submitted 2013-02-13; First posted 2013-02-28 (Estimated); Results first posted 2016-09-09 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Transplantation; Immunosuppression; Drug Interaction
Keywords: immunosuppressive medication; mycophenolic acid; interaction; proton pump inhibitor; pantoprazole; renal transplant patients; pharmacokinetics; pharmacodynamics; bioavailability
MeSH Terms: interventions — Mycophenolic Acid; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mycophenolate mofetil (C) (Active Comparator): Mycophenolate mofetil (C) b.i.d. every 12 hours for 2 weeks.
  Interventions: Drug: Mycophenolate mofetil
- Mycophenolate mofetil+Pantoprazole (C+P) (Other): Mycophenolate mofetil b.i.d and Pantoprazole o.m. for 2 weeks.
  Interventions: Drug: Pantoprazole; Drug: Mycophenolate mofetil
- Mycophenolate sodium (M) (Other): Mycophenolate sodium (M) b.i.d. every 12 hours for 2 weeks.
  Interventions: Drug: Mycophenolate sodium
- Mycophenolate sodium+Pantoprazole (M+P) (Other): Mycophenolate mofetil b.i.d and Pantoprazole 40mg o.m. for 2 weeks.
  Interventions: Drug: Mycophenolate sodium; Drug: Pantoprazole

INTERVENTIONS:
Drug: Mycophenolate sodium — Daily dose: 720mg, 1080mg, 1440mg. Application alone or together with Pantozol®.
  Other Names: Myfortic®
  Arms: Mycophenolate sodium (M); Mycophenolate sodium+Pantoprazole (M+P)
Drug: Pantoprazole — Daily dose: 40mg. Application together with CellCept® or Myfortic® .
  Other Names: Pantozol®
  Arms: Mycophenolate mofetil+Pantoprazole (C+P); Mycophenolate sodium+Pantoprazole (M+P)
Drug: Mycophenolate mofetil — Daily dose: 1000mg, 1500mg, 2000mg. Application alone or with Pantozol® .
  Other Names: Cellcept®
  Arms: Mycophenolate mofetil (C); Mycophenolate mofetil+Pantoprazole (C+P)

SUMMARY:
The objective of this pharmacokinetic study is to examine a possible drug-drug interaction of Pantoprazole on the bioavailability mycophenolic acid.

DETAILED DESCRIPTION:
It is a randomized open-label 4-sequence 4-period pharmacokinetic cross-over study. The objective of the pharmacokinetic study is to examine a drug-drug interaction of pantoprazole on the bioavailability mycophenolic acid administered as either mycophenolate mofetil (Cellcept(R) or mycophenolate Sodium; EC-MPS (Myfortic (R) in stable renal allograft recipients under maintenance immunosuppressive therapy (cyclosporine +/- low dose glucocorticoids).

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years old
* patients who are on stable immunosuppressive therapy for at least one month with ciclosporin, EC-MPS or MMF +/- corticosteroids
* renal transplantation, at least 6 months prior study inclusion
* suitable and willing to switch treatment according to the study plan
* women of childbearing potential must have a negative serum pregnancy test before study start and effective contraception must be used (method with PEARL index <1%)

Exclusion Criteria:

* patients with renal function <30ml/min (estimated by Cockcroft Gault formula)
* patients who are not on stable treatment with enzyme inductors or enzyme inhibitors for <1 month before study entry
* patients who take medication which is known for interfering with MPA absorption for <1 month before study entry
* known anamnestic hypersensitivity to one of the investigational products or drugs with similar chemical structure and to other components of the investigational products, respectively
* patients on treatment with clopidogrel
* acute rejection < 1 month before study inclusion
* patients who are HIV positive, hepatitis C virus (HCV) positive, HBsAg positive
* patients with gastrointestinal disorders which could affect resorption
* pregnancy and/or lactation
* drug or alcohol abuse in patient's history
* patients with history of psychological illness or condition, which might interfere with the ability to understand the requirements, consequences, possible outcome of the study and patients who are not willing to give valid informed consent
* patients with insufficient co-operation with the clinical investigator (e.g. suspicion of non-compliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klemens Budde, Prof Dr, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Hospital Campus Mitte, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment lastet between January 2012 - March 2013.
Groups:
- Sequence A: 1. st period: Mycophenolate mofetil (MMF) tablet (500, 750 or 1000mg) b.i.d. every 12 hours for 10-14d.
  2. nd period: Mycophenolate sodium (EC-MPS) tablet (720, 1080, 1440) b.i.d. every 12 hours for 10-14d.
  3. rd period: Mycophenolate sodium (EC-MPS) tablet (720, 1080, 1440) b.i.d. every 12 hours for 10-14d. Pantoprazole 40mg tablet (PAN) each for 10-14d.
  4. th period: Mycophenolate mofetil (MMF) tablet (500, 750 or 1000mg) b.i.d. every 12 hours for 10-14d. Pantoprazole 40mg tablet (PAN) each for 10-14d.
- Sequence B: 1. st period: Mycophenolate sodium (EC-MPS) tablet (720, 1080, 1440) b.i.d. every 12 hours for 10-14d.
  2. nd period: Mycophenolate sodium (EC-MPS) tablet (720, 1080, 1440) b.i.d. every 12 hours for 10-14d. Pantoprazole 40mg tablet (PAN) each for 10-14d.
  3. rd period: Mycophenolate mofetil (MMF) tablet (500, 750 or 1000mg) b.i.d. every 12 hours for 10-14d. Pantoprazole 40mg tablet (PAN) each for 10-14d.
  4. th period: Mycophenolate mofetil (MMF) tablet (500, 750 or 1000mg) b.i.d. every 12 hours for 10-14d.
- Sequence C: 1. st period: Mycophenolate sodium (EC-MPS) tablet (720, 1080, 1440) b.i.d. every 12 hours for 10-14d. Pantoprazole 40mg tablet (PAN) each for 10-14d.
  2. nd period: Mycophenolate mofetil (MMF) tablet (500, 750 or 1000mg) b.i.d. every 12 hours for 10-14d. Pantoprazole 40mg tablet (PAN) each for 10-14d.
  3. rd period: Mycophenolate mofetil (MMF) tablet (500, 750 or 1000mg) b.i.d. every 12 hours for 10-14d.
  4. th period: Mycophenolate sodium (EC-MPS) tablet (720, 1080, 1440) b.i.d. every 12 hours for 10-14d.
- Sequence D: 1. st period: Mycophenolate mofetil (MMF) tablet (500, 750 or 1000mg) b.i.d. every 12 hours for 10-14d. Pantoprazole 40mg tablet (PAN) each for 10-14d.
  2. nd period: Mycophenolate mofetil (MMF) tablet (500, 750 or 1000mg) b.i.d. every 12 hours for 10-14d.
  3. rd period: Mycophenolate sodium (EC-MPS) tablet (720, 1080, 1440) b.i.d. every 12 hours for 10-14d.
  4. th period: Mycophenolate sodium (EC-MPS) tablet (720, 1080, 1440) b.i.d. every 12 hours for 10-14d. Pantoprazole 40mg tablet (PAN) each for 10-14d.
Period: Period 1
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started | 5 (Each period lasted 10-14 weeks) | 5 | 5 | 5
Completed | 5 | 4 | 5 | 5
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started | 5 | 4 | 5 | 5
Completed | 4 | 4 | 5 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started | 4 | 4 | 5 | 5
Completed | 4 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started | 4 | 4 | 5 | 5
Completed | 4 | 4 | 4 | 5
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: y] — Age at transplantation
  y | 59 (12) | 42 (14) | 33 (17) | 43 (14) | 44 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4 | 8
  Male | 3 | 3 | 5 | 1 | 12
Age at study enrollment [Mean (Standard Deviation); unit: years] | 63 (11) | 46 (16) | 44 (15) | 51 (19) | 51 (16)

OUTCOME MEASURES:

1. Primary Outcome: Dose-normalized AUC of Mycophenolic Acid
Description: Bioavailability (12h AUC) of mycophenolic acid in renal transplant patients after administration of MMF+/-PAN and EC-MPS+/-PAN
  For evaluation of pharmacokinetic and pharmacodynamic parameters blood will be collected before, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h after drug intake.
Time Frame: Study duration for each patient: 2 months. After 10-14 days of drug intake blood samples for PK/PD analysis will be collected. On the next day new treatment starts. There are 4 study visits at the study center. Duration will be approximately 12hours
Measure: Mean (Standard Deviation); unit: mg*h/L
Groups:
- Mycophenolate Mofetil (MMF): Mycophenolate mofetil (MMF) tablet twice a day every 12 hours for two weeks.
  Mycophenolate mofetil daily dose: 1000mg, 1500mg, 2000mg.
- MMF+PAN: Mycophenolate mofetil (MMF) tablet twice a day every 12 hours for two weeks.
  Mycophenolate mofetil daily dose: 1000mg, 1500mg, 2000mg.
  Pantoprazole daily dose: 40mg once in the morning together with Mycophenolate mofetil.
  Pantoprazole tablet (PAN) once a day in the morning for two weeks.
- EC-MPS: Mycophenolate sodium (EC-MPS) tablet twice a day every 12 hours for two weeks.
  Mycophenolate sodium daily dose: 720mg, 1080mg, 1440mg.
- EC-MPS + PAN: Mycophenolate sodium (EC-MPS) tablet twice a day every 12 hours for two weeks.
  Mycophenolate sodium daily dose: 720mg, 1080mg, 1440mg.
  Pantoprazole daily dose: 40mg once in the morning together with Mycophenolate sodium.
  Pantoprazole tablet (PAN) once a day in the morning for two weeks.
Arm/Group | Mycophenolate Mofetil (MMF) | MMF+PAN | EC-MPS | EC-MPS + PAN
Number analyzed (Participants) | 17 | 17 | 17 | 17
mg*h/L | 41 (18) | 38 (18) | 43 (19) | 46 (18)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at every study visit. No follow up data.
Groups:
- MMF + PAN: Mycophenolate mofetil (MMF) tablet twice a day every 12 hours for two weeks.
  Mycophenolate mofetil daily dose: 1000mg, 1500mg, 2000mg.
  Pantoprazole daily dose: 40mg once in the morning together with Mycophenolate mofetil.
  Pantoprazole tablet (PAN) once a day in the morning for two weeks.
Arm/Group | Mycophenolate Mofetil (MMF) | MMF + PAN | EC-MPS | EC-MPS + PAN
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 4/19 | 3/18 | 2/18 | 2/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (MMF) (N=19) | MMF + PAN (N=18) | EC-MPS (N=18) | EC-MPS + PAN (N=18)
Noro virus infection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (MMF) (N=19) | MMF + PAN (N=18) | EC-MPS (N=18) | EC-MPS + PAN (N=18)
Common cold (Immune system disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes